CLINICAL TRIAL: NCT00531310
Title: A Pilot Study of Reduced Intensity Allogeneic Stem Cell Transplantation in Patients With Chronic Myeloid Leukemia (CML) and Adoptive Cellular Immunotherapy Only in Patients With Persistent Disease and Matched Family Donors
Brief Title: Reduced Intensity AlloSCT in(CML) With Persistent Disease
Acronym: CML
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Columbia University (Other)
Responsible Party: Mitchell Cairo, MD, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAA8191; CHNY-01-505 (Other: CU)
Record Dates: First submitted 2007-09-15; First posted 2007-09-18 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Myeloid Leukemia
Keywords: CML; allogeneic SCT; matched family donor; unrelated donor; cord blood donor; persistent disease
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Busulfan; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Matched Family Donor (Experimental): Matched Family Donor
  Interventions: Drug: Reduced Intensity Conditioning, Busulfan and Fludarabine
- Unrelated Donor (Experimental): Unrelated Donor Transplant/ Cord Blood Transplant
  Interventions: Drug: Reduced Intensity Conditioning, Busulfan and Fludarabine

INTERVENTIONS:
Drug: Reduced Intensity Conditioning, Busulfan and Fludarabine — Busulfan and Fludarabine
  Other Names: RIC

SUMMARY:
CML, a malignant disorder of stem cells, is characterized by increases in both immature and mature myeloid, erythroid, and lymphoid cells, as well as platelets in the peripheral blood. The cytogenetic hallmark of CML is the Philadelphia(Ph)chromosome found in the malignant cells of 95% of patients. CML comprises 7-20% of all leukemias with an overall incidence in the general population estimated at 1 to 2 per 100,000. The peak incidence occurs in the fifth decade, however, all age groups, including children, are affected. The only reported environmental risk factor is exposure to excessive ionizing radiation that is documented in only a very small percentage of patients. Clinically, CML is characterized by an initial chronic phase in which patients may report mild constitutional symptoms; however, 40-50% are asymptomatic and are diagnosed based upon abnormal blood counts discovered during a routine examination. The chronic phase typically lasts three to five years, and is followed by an accelerated phase distinguished by progressive systemic symptoms, an increasing resistance to conventional chemotherapy, and a rise in the peripheral blood and bone marrow blast count. This evolves rapidly into a blastic crisis characterized by immature cells resembling the blasts characteristic of acute leukemia. The presence of 30% or more blastic cells in the blood or marrow is diagnostic of this final blastic phase which is typically fatal within 3 to 6 months.

The primary treatment options for CML have traditionally been monotherapy with either busulfan or hydroxyurea. Both agents are able to control the clinical symptoms associated with CML, as well as induce hematological remissions in 80% of chronic phase patients. However, complete cytogenetic remissions with either agent are rare, and neither is able to prevent eventual progression to the terminal blastic phase; therefore, these therapies can only be considered palliative.

The primary purpose of this clinical research trial is to study the feasibility of a reduced intensity allogenic transplant for CML. This study will also determine the side effects as well as the response rate.

DETAILED DESCRIPTION:
Further study details will be provided by Columbia University, Division of Pediatric Blood and Marrow Transplantation.

STUDY DESIGN:

Patients less than 30 years of age with CML in 1st or 2nd chronic phase or 1st accelerated phase and a matched related donor, an unrelated cord blood donor, or an unrelated adult donor, will receive 6 days of IV Fludarabine, 4 doses of IV Busulfex, and 5 doses of Alemtuzumab. Patients with persistant RT-PCR positive BCR-Abl and/or Philadelphia chromosome positivity by cytogentics after Day + 100 and a matched related donor would receive DLIx1. If still BCR-Abl or Philadelphia chromosome positive at Day +180 and a matched related donor, patients would receive a second dose of DLI. All patients will receive STI-571 (Gleevec) after hematological reconstitution. Studies for immune reconstitution, chimersim, and MRD will be performed postt AlloSCT.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patient must be less than 30 years of age.
* Consent: Patient or the patient's legally authorized guardian must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects), and must sign an informed consent in accordance with the institutional policies approved by the U.S. Department of Health and Human Services.
* Organ Function: Patient must have adequate organ function as below Adequate renal function defined as:Serum creatinine 1.5 x normal, or Creatinine clearance or radioisotope GFR > 40 ml/min/m2 or >60 ml/min/1.73 m2 or an equivalent GFR as determined by the institutional normal range
* Adequate liver function defined as:Total bilirubin < 2.5 x normal; or SGOT (AST) or SGPT (ALT) < 5.0 x normal
* Adequate cardiac function defined as:

  * Shortening fraction of >25% by echocardiogram, or
  * Ejection fraction of >40% by radionuclide angiogram or echocardiogram
* Adequate pulmonary function defined as:

  -DLCO >40% by pulmonary function test For children who are uncooperative, no evidence of dyspnea at rest,no exercise intolerance, and a pulse oximetry >94% in room air.
* Disease Status

  * Patients with CML with either of the following:
  * Patients in 1st or 2nd chronic phase
  * Patients in 1st or 2nd accelerated phase

Exclusion Criteria:

* Patient in blast crisis
* Patient in 3rd or greater chronic phase
* Patient in 3rd or greater accelerated phase

  * women that are pregnant are ineligible

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2003-01; Primary Completion 2007-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To determine the toxicity associated with reduced intensity therapy and allogeneic SCT in selected patients with CML. | Until Study End

CONTACTS AND LOCATIONS:
Overall Officials: Mtchell S Cairo, MD, Principal Investigator — Columbia University
Locations (1):
- Morgan Stanley Children's Hospital of NYP, New York, New York, United States